CLINICAL TRIAL: NCT04969549
Title: Use of Functional Neuroimaging Biomarkers as Early Predictors of Response to Theta-burst Stimulation Treatment in Depression
Brief Title: Response Predictors of Theta-burst Stimulation for Depression
Acronym: TBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Academy of Medical Sciences, UK (Other)
Responsible Party: Principal Investigator, Andre R Brunoni, Associate Professor of the Medical School of the University of Sao Paulo (FMUSP), Principal Investigator, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 43768721.4.0000.0068; NAFR12\1010 (Other Grant/Funding Number: Academy of Medical Sciences UK)
Record Dates: First submitted 2021-07-16; First posted 2021-07-20 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Depression
Keywords: depression; TBS; fMRI; response predictors
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Active TBS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Theta-burst stimulation (TBS) (Other): Receive active iTBS, 1800 pulses, 100% MT over dlPFC.
  Interventions: Other: Theta burst stimulation

INTERVENTIONS:
Other: Theta burst stimulation — It consists of 20 sessions of iTBS over the dlPFC.
  Other Names: TBS

SUMMARY:
The study consists of an open label trial designed to treat adult depression with TBS. Our aim is to build capacity in neuroimaging analyses by performing magnetic resonance imaging (MRI) assessments at baseline and after 7-10 days of treatment onset in 70 patients. The scientific goal is to test a hypothesis about treatment action: that TBS will reduce negative bias (which causally maintains negative mood) after 1 week of treatment, and patients who show this neurocognitive change will be the ones who go on to respond clinically after 6 weeks.

DETAILED DESCRIPTION:
Depressive disorders are among the leading causes of incapacity and disability worldwide. The burden of depression is expected to increase and is associated with negative impact on clinical conditions and physical and cognitive abilities. Given the limited efficacy of antidepressant drugs, novel treatments such as theta-burst brain stimulation (TBS), a form of repetitive transcranial magnetic stimulation (rTMS), are being developed. However, to further advance the field towards treatment personalisation, increasing understanding of TBS antidepressant mechanisms and identifying treatment responders are important issues. Moreover, no studies have used neuroimaging in TBS trials in depression yet. Our group in Brazil is a leading brain stimulation centre, although neuroimaging expertise is lacking. We will conduct an open label trial designed to treat adult depression with TBS. Our aim is to build capacity in neuroimaging analyses by performing magnetic resonance imaging (MRI) assessments at baseline and after 7-10 days of treatment onset in 70 patients. The scientific goal is to test a hypothesis about treatment action: that TBS will reduce negative bias (which causally maintains negative mood) after 1 week of treatment, and patients who show this neurocognitive change will be the ones who go on to respond clinically after 6 weeks. Scientifically, this proposal and its outcomes will help advance towards next-generation precision brain stimulation, by incorporating cognitive/neuroimaging readouts that inform about mechanism and individual response.

ELIGIBILITY:
Inclusion Criteria: participants aged from 18 to 65 years, with HDRS score ≥ 14, with MDD confirmed by MINI structured interview.

-

Exclusion Criteria: other mental disorders (alcohol or other substance dependence, bipolar disorder, psychotic disorders or dementia), severe clinical or neurological disorders, suicidal ideation, presence of psychotic symptoms, severe depression characterized by HDRS score > 28, manic symptoms characterized by score > 8 in the Young Mania Rating Scale. In addition, patients with specific contraindications to magnetic stimulation or magnetic resonance imaging will be excluded, such as having any metallic implants, epilepsy or any electronic component in the head.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale scores (17-item version) | Week 0 (baseline) and Week 6
  Clinician-administered depression assessment scale. Score range = 0 - 52 (higher scores mean worse outcome).

SECONDARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale scores (MADRS) | Week 0 (baseline) and Week 6
  Clinician-administered depression assessment scale. Score range = 0 - 60 (higher scores mean worse outcome).
Change in Young Mania Rating Scale (YMRS) scores | Week 0 (baseline) and Week 6
  Clinician-administered scale that measures hypomania/mania symptoms. Score range = 0 - 60 (higher scores mean worse outcome).
Facial Expression Recognition Test (FERT) | Week 0 (baseline) and Week 2.
  Cognitive test used to detect emotional bias.
Change in Positive and Negative Affect Schedule scores (PANAS) | Week 0 (baseline) and Week 6
  Self-report questionnaire to measure both positive and negative affect. Positive Affect Score: scores can range from 10 - 50, with higher scores representing higher levels of positive affect (better outcome). Negative Affect Score: scores can range from 10 - 50, with higher scores representing higher levels of negative affect (worse outcome).
Change in State-Trait Anxiety Inventory scores (STAI-T and STAI-S) | Week 0 (baseline) and Week 6
  Self-report measures of state and trait anxiety. The range of possible scores for each subscale (STAI-T and STAI-S) varies from a minimum score of 20 to a maximum score of 80, with higher scores meaning worse outcome.
Change in functional and structural neuroimaging exam | baseline and after two weeks
  Neuroimaging exam used to measure both functional and structural aspects of the brain as possible predictors of clinical response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Andre R Brunoni, MD, PhD, Principal Investigator — FACULDADE DE MEDICINA DA USP
Locations (1):
- Instituto de Psiquiatria, São Paulo, São Paulo, Brazil